CLINICAL TRIAL: NCT06031519
Title: Impact of Percutaneous Intramyocardial Septal Radiofrequency Ablation in Obstructive Hypertrophic Cardiomyopathy on Arrhythmias
Brief Title: Impact of Liwen Procedure in Obstructive Hypertrophic Cardiomyopathy on Arrhythmias
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Liu Liwen, Director, Xijing Hospital
Other Study IDs: KY-20232259-C-1
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Hypertrophic Cardiomyopathy; Arrhythmia
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypertrophic Obstructive Cardiomyopathy Patients underwent Liwen Procedure
  Interventions: Procedure: Percutaneous Intramyocardial Septal Radiofrequency Ablation for hypertrophic obstructive cardiomyopathy (Liwen Procedure)

INTERVENTIONS:
Procedure: Percutaneous Intramyocardial Septal Radiofrequency Ablation for hypertrophic obstructive cardiomyopathy (Liwen Procedure) — Under transthoracic echocardiography (TTE) guidance, the puncture site is positioned at the apex. A guiding line is applied along the septal long axis and the radiofrequency ablation electrode needle(17G, Cool-tip™ RF Ablation System and Switching Controller; Medtronic, Minneapolis, MN, USA) pierced towards the hypertrophic anterior interventricular septum (AIVS) 8-10 mm from the subaortic valve. Each ablation lasts up to 12 min, and the ablation power gradually increases from 30-40W. Then, the ablation needle is withdrawn 10 mm to prepare for the next application. Overall, 3-4 applications are performed in each patient. The ablation creates an area of thermal coagulative myocardial necrosis that appears as a hyperechogenic reflection detected by TTE. If deemed necessary, we repeat the procedure at the posterior interventricular septum (PIVS).

SUMMARY:
The goal of this observational study is to learn about the occurrence of various arrhythmias ( tachyarrhythmia and bradyarrhythmia ) during or after Percutaneous Intramyocardial Septal Radiofrequency Ablation. The main questions it aims to answer are:

* To investigate the occurrence of various arrhythmias ( tachyarrhythmia and bradyarrhythmia ) during procedure and its relationship with clinical characteristics and procedural parameters
* To analyze the changes of 12-lead electrocardiogram and 24-hour dynamic electrocardiogram before and after Percutaneous Intramyocardial Septal Radiofrequency Ablation and their relationships with clinical characteristics and procedural parameters

ELIGIBILITY:
Inclusion Criteria:

1. Subject with symptoms that limit daily activities (New York Heart Association functional class >II, exercise-induced syncope) despite adequate medical treatment or when medical treatment is not tolerated
2. Subject with a peak LVOT gradient≥50 mm Hg
3. Subject volunteers for the Liwen procedure and received the procedure at the Hypertrophic Cardiomyopathy Center of Xijing Hospital.

Exclusion Criteria:

1. Subject with a peak instantaneous Doppler LVOT gradient of <50 mm Hg
2. Subject with an indication for septal reduction therapy and other lesions requiring surgical intervention (e.g., mitral valve repair/replacement and papillary muscle intervention)
3. Subject has end-stage heart failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are diagnosed with obstructive HCM and with drug-refractory symptoms underwent Liwen Procedure in Xijing Hospital from 2016 to 2023.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
All-cause and cardiovascular mortality | From date of procedure until the date of first occurrence of outcome, assessed up to 1 years
  All-cause and cardiovascular mortality (defined as sudden cardiac death, Heart Failure-related death, and heart transplant) were the primary outcomes.

SECONDARY OUTCOMES:
Ventricular tacharrhythmia composite outcome | From date of procedure until the date of first occurrence of outcome, assessed up to 1 years
  Unexplained syncope, resuscitated cardiac arrests, or appropriate implantable cardioverter-defibrillator charge.
Arrhythmia | From date of procedure until the date of first occurrence of outcome, assessed up to 1 years
  Complete heart block, new permanent pacemaker implantation, non-sustained ventricular tachycardia, sustained ventricular tachycardia, left bundle branch block, right bundle branch block, premature ventricular contractions burden more than 10% monitored by Holter.

CONTACTS AND LOCATIONS:
Locations (1):
- Ultrasound Medicine Department of Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China